CLINICAL TRIAL: NCT04379765
Title: Long-term Follow-up of Conservative and Surgical Treatment Results of Patients With Lumbar Spinal Stenosis
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Medical Doctor in Physical Medicine and Rehabilitation, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2373
Record Dates: First submitted 2020-03-19; First posted 2020-05-07 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spinal Stenosis; Rehabilitation; Surgery; Exercise
MeSH Terms: conditions — Spinal Stenosis; Motor Activity | interventions — Exercise; Physical Therapy Modalities; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grup 1: Exercise and physical therapy programme: 30 patients with lumbar spinal stenosis will receive hot pack, transcutaneous electrical nerve stimulation and deep warming as a physical therapy modality , and lumber flexion and strengthening exercises were performed for 7 times/week for 3 weeks.
  Interventions: Behavioral: Exercise and physical therapy
- Grup 2: Surgical procedure programme: 30 patients with lumbar spinal stenosis underwent decompression operation of the relevant level.

INTERVENTIONS:
Behavioral: Exercise and physical therapy — Decompression operation
  Other Names: Surgery
  Groups: Grup 1: Exercise and physical therapy programme

SUMMARY:
Total of 60 patients with a diagnosis of spinal stenosis is planned for 30 patients, with physical therapy modeling and exercise, and 30 patients with surgical treatment. Patients will be evaluated by the same physician 5 times, before early primary treatment, 1st month, 3rd month, 6th month and 12th month after treatment.

DETAILED DESCRIPTION:
Patients between 40-85 years old who are hospitalized and treated with the diagnosis of LSS in Physical Medicine and rehabilitation, Orthopedics and Neurosurgery Clinics will be included in the study. The diagnosis of LSS will be made by MR and / or CT and neurogenic claudication history.

Total of 60 patients with a diagnosis of spinal stenosis is planned for 30 patients, with physical therapy modeling and exercise, and 30 patients with surgical treatment, and the duration of the study is considered to be 24 months. Patients will be evaluated by the same physician 5 times, before early primary treatment, 1st month, 3rd month, 6th month and 12th month after treatment.

Clinical evaluation will be done by the same physician. In patients with spinal stenosis, pain (movement, rest, night) VAS, functional status walking distance and ILBDI (Istanbul waist pain disability index) inquiry form, Nottingham Extended Life Profile will be used.

ELIGIBILITY:
Inclusion Criteria:

1. To be between 40-85 years old
2. Defining neurogenic claudication in patient anamnesis
3. Diagnosis of lumbar stenosis in MR and / or CT imaging
4. The duration of the symptom should be at least 4 weeks
5. Other causes of low back pain have been ruled out

Exclusion Criteria:

1. Having had lumbar surgery before
2. Physical therapy for lumbar spinal stenosis less than 3 months ago
3. Any lumbar injection has been applied before
4. Patients with inflammatory low back pain
5. Patients with spinal stenosis due to spondylolysis and / or spondylolisthesis
6. Patients with a history of trauma and suspected Vertebral fracture

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: It is planned to take 60 patients with a diagnosis of spinal stenosis to perform physical therapy models and exercise for 30 patients and surgical treatment for 30 patients. Patients between the ages of 40-85 will be admitted and no difference will be made in terms of gender. The child patient will not be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation VAS (visual analog scale) for pain assessment | 1st month
  Clinical evaluation will be done by the same physician. In patients with spinal stenosis, VAS (visual analog scale) for pain assessment will be used.
Clinical Evaluation 2 functional status walking distance | 1st month
  In patients with spinal stenosis, functional status walking distance will be used.
Clinical Evaluation 3 Istanbul waist pain disability index | 1st month
  In patients with spinal stenosis, ILBDI (Istanbul waist pain disability index) form will be used.
Clinical Evaluation 4 Nottingham Extended Life Profile | 1st month
  In patients with spinal stenosis, Nottingham Extended Life Profile will be used.

SECONDARY OUTCOMES:
Clinical Evaluation 5 | 12th month
  In patients with spinal stenosis, VAS will be used in 3rd , 6th and 12th month.
Clinical Evaluation 6 | 12th month
  In patients with spinal stenosis, functional status walking distance will be used in 3rd , 6th and 12th month.
Clinical Evaluation 7 | 12th month
  In patients with spinal stenosis, ILBDI (Istanbul waist pain disability index) form will be used in 3rd , 6th and 12th month.
Clinical Evaluation 8 | 12th month
  In patients with spinal stenosis, Nottingham Extended Life Profile will be used in 3rd , 6th and 12th month.

CONTACTS AND LOCATIONS:
Overall Officials: Figen Yılmaz, Prof. Dr., Principal Investigator — Şişli Hamidiye Etfal Research and Training Hospital
Locations (1):
- Science Health University Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tsubosaka M, Kaneyama S, Yano T, Kasahara K, Kanemura A, Takabatake M, Hirata H, Sumi M. The factors of deterioration in long-term clinical course of lumbar spinal canal stenosis after successful conservative treatment. J Orthop Surg Res. 2018 Sep 18;13(1):239. doi: 10.1186/s13018-018-0947-2. PMID 30227869